CLINICAL TRIAL: NCT01530087
Title: Peristomal Skin Irritation: A Preliminary Evaluation of the CASTLE Barrier Prototype for People With Intestinal Stomas
Brief Title: Preliminary Evaluation of CASTLE Barrier Prototype UK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability of site to recruit/enroll target population
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4518-O; CIV-GB-11-07-001241 (Registry Identifier: Eudamed)
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-09

CONDITIONS: Peristomal Skin Complication
Keywords: colostomy; ileostomy; irritant dermatitis; two piece barrier
MeSH Terms: conditions — Dermatitis, Irritant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): CASTLE Barrier
  Interventions: Device: CASTLE barrier

INTERVENTIONS:
Device: CASTLE barrier — Prototype barrier to be used in place of current two piece device

SUMMARY:
The purpose of this study is to provide preliminary assessment of the safety and performance of a novel barrier formulation (CASTLE) in a small population of subjects with irritated peristomal skin.

DETAILED DESCRIPTION:
This is a single-site, unblinded, historically controlled, first use in humans study of a stoma barrier with a new formulation. Approximately 34 subjects who are currently using a 2-piece tape bordered product and able and willing to wear a product will be enrolled. Each participant is provided with one box containing 20 of the test barriers to be used consecutively according to their normal routine. Each participant is also provided with a box containing 30 pouches selected to most closely resemble their current product. Participants are asked to record the time of application and time of removal of each test barrier and their assessment of relevant characteristics for each test barrier. A clinical evaluation of the peristomal skin is conducted at study entry, at approximately mid way through the study and again at its conclusion. Photographs are taken of the peristomal skin at each visit using a digital camera. Individual participation in terms of wearing the barrier is for 30 days or until the test barrier has been used up, whichever comes first. The study is comprised of 3 visits, an enrolment visit, a mid-study visit and a completion visit and a phone call at approximately day 7.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* has colostomy or ileostomy
* current uses two piece tape bordered barrier
* has mild to moderate peristomal skin irritation
* cares for their stoma independently in the community
* at least 3 months post-operative
* provides informed consent

Exclusion Criteria:

* has fistula on or near stoma
* has been involved in stoma care study in the last 30 days
* is pregnant or lactating (determined by interview only)
* has existing medical condition that would compromise their participation or follow-up
* currently uses convex ostomy products, paste and/or rings
* is allergic to test barrier components
* is undergoing chemo- or radiotherapy that may affect the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Murahata, PhD, Study Director — Hollister Incorporated
Locations (1):
- York Teaching Hospital, York, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Ileostomy or Colostomy: CASTLE Barrier ostomy device
  CASTLE barrier: Prototype barrier to be used in place of current two piece device
Period: Overall Study
Arm/Group | Subjects With Ileostomy or Colostomy
Started | 3
Completed | 1
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Ileostomy or Colostomy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Peristomal Skin Condition
Description: mean irritation score using a categorical scale with range of 1(normal) to 5(eroded or heaemorrhagic dermatitis)
Time Frame: 1 - 30 days
Population: Study was stopped due to inability to inability to enroll. No data are available for any outcome measures.
Groups:
- Treatment: CASTLE Barrier: Prototype barrier used in place of previous two piece device
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Security
Description: wear time leakage barrier erosion
Time Frame: 30 days
Population: Study was stopped ; no data are available
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Subjects With Ileostomy or Colostomy
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other